CLINICAL TRIAL: NCT06469541
Title: Clinical Outcomes After Implantation of a Monofocal Hydrophobic IOL, Bi-Flex 877PAY With POB-MA Preloaded Injector: Visual Outcomes, Refractive Stability, Safety Features, YAG Capsulotomy Rate. (Retrospective Review)
Brief Title: Clinical Outcomes After Implantation of a Monofocal Hydrophobic IOL, Bi-Flex 877PAY With POB-MA Preloaded Injector
Status: Completed | Type: Observational
Sponsor: Medicontur Medical Engineering Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: M-877PAY-UK-2008
Record Dates: First submitted 2023-05-31; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2023-04

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of our investigation is to retrospectively assess visual outcomes, refractive stability, safety features of the lens and the incidence of developing PCO (posterior capsular opacification) in a 12-month period following mono- or bilateral implantation of the hydrophobic acrylic monofocal IOL, Bi-Flex 877PAY (Medicontur).

DETAILED DESCRIPTION:
The purpose of our investigation is to retrospectively assess visual outcomes, refractive stability, safety features of the lens and the incidence of developing PCO (posterior capsular opacification) in a 12-month period following mono- or bilateral implantation of the hydrophobic acrylic monofocal IOL, Bi-Flex 877PAY (Medicontur).

* Primary objective:

  o To evaluate the monocular Uncorrected Distance Visual Acuity (UCDVA) 1 year after IOL implantation
* Secondary objectives:

  * To evaluate the spherical equivalent refraction one month postoperatively.
  * To evaluate level of astigmatism one month postoperatively.
  * To evaluate the Uncorrected Distance Visual Acuity (UDVA) monocular at 1 day, 1 month and 6 months after IOL implantation
  * To evaluate the Best Corrected Distance Visual Acuity (CDVA) monocular at 1 month, 6 months and 1 year after IOL implantation
  * To evaluate safety features of the lens
  * To evaluate PCO development, Nd:YAG capsulotomy rate

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients who underwent cataract surgery in one or both eyes and who were implanted with Bi-Flex 877PAY IOL mono- or bilaterally.
2. Patients with regular post-operative visits over 12 months period after surgery.
3. Patients of any age above 18 years and any medical history who are eligible according the investigator's decision.

Exclusion Criteria:

1. preoperative corneal astigmatism > 1.5 D
2. uncontrolled diabetic retinopathy
3. iris neovascularisation
4. serious intraoperative complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The enrolled subjects will be the patients who underwent cataract surgery in one or both eyes and who were implanted with Bi-Flex 877PAY IOL mono- or bilaterally. For evaluation of records consecutive implanted patients with regular post-operative visits over a 12 months period will be included.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-04-11 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Primary objective | 12 months after IOL implantation
  To evaluate the monocular Uncorrected Distance Visual Acuity (UCDVA) 1 year after IOL implantation

SECONDARY OUTCOMES:
Secondary onjective | 12 months after IOL implantation
  To evaluate the spherical equivalent refraction one month postoperatively. To evaluate level of astigmatism one month postoperatively. To evaluate the Uncorrected Distance Visual Acuity (UDVA) monocular at 1 day, 1 month and 6 months after IOL implantation To evaluate the Best Corrected Distance Visual Acuity (CDVA) monocular at 1 month, 6 months and 1 year after IOL implantation To evaluate safety features of the lens To evaluate PCO development, Nd:YAG capsulotomy rate

CONTACTS AND LOCATIONS:
Overall Officials: Sathish Srinivasan, Prof., Principal Investigator — NHS Ayrshire and Arran
Locations (1):
- NHS Ayrshire and Arran, Ayr, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No